CLINICAL TRIAL: NCT03328572
Title: Clinical Performance and Patient Satisfaction of Cerasmart Versus Lithium Disilicate (E-max) Endocrowns of Endodontically Treated Molar Teeth
Brief Title: Clinical Performance and Patient Satisfaction of Cerasmart Versus Lithium Disilicate (E-max) Endocrowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moustafa Elbehairy, PhD Student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: CEBD-CU-2017-10-27
Record Dates: First submitted 2017-10-23; First posted 2017-11-01 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- E-max Endocrowns (Active Comparator): all patients in this arm will receive e-max endocrowns
  Interventions: Other: E-max Endocrown
- Cerasmart Endocrowns (Experimental): all patients in this arm will receive Cerasmart endocrowns
  Interventions: Other: Cerasmart Endocrown

INTERVENTIONS:
Other: E-max Endocrown — Endocrown preparation
  Arms: E-max Endocrowns
Other: Cerasmart Endocrown — Endocrown preparation
  Arms: Cerasmart Endocrowns

SUMMARY:
1. RATIONALE All-ceramic endocrowns are bonded to the tooth using adhesive resins creating strong bonds to the tooth structure resulting in strengthening effect and reducing the need for post and core. various CAD/CAM materials can be used for the fabrication of endocrowns including lithium-disilicate reinforced glass-ceramics, feldspathic ceramics, in ceram alumina and in ceram spinell as well as hybrid ceramics and composites.

   Fewer data are available on the clinical performance of the different materials used for endocrowns. With the rapid innovation in the dental restorative materials clinicians are sometimes confused when selecting the best restorative material to restore an endodontically treated tooth with an endocrown. This is due to lack of data with regard to clinical performance of these restorations as well as the degree of patient satisfaction.
2. OBJECTIVES P= Endodontically treated teeth indicated for endocrown I1= Feldspathic endocrown I2= Hybrid endocrown C= IPS e.max Endocrown O= Clinical performance

Research question In patients with endodontically treated teeth requiring endocrown restorations, what are the clinical performance and the level of patient satisfaction of cerasmart endocrown versus lithium disilicate (e-max) ceramic endocrowns?

DETAILED DESCRIPTION:
Administrative information

1. Title: Clinical performance and patient satisfaction of cerasmart versus lithium disilicate (e-max) endocrowns of endodontically treated teeth (Randomized Controlled Clinical trial) 2. Trial registration: This study will be registered on Clinicaltrials.gov. 3. Protocol version: Version (1). 4. Funding: The trial is totally self-funded whether on a financial or a non-financial basis. Department of fixed prosthodontics, Faculty of Oral and Dental Medicine, Cairo University, provides equipment units and some consumables.

5. Roles and responsibilities 5.a. Name: Moustafa Maher Moustafa Elbehairy (E.M). Rule: (Main researcher*)

*Responsible for all clinical procedure in this clinical trial and measuring different outcomes for each group.

Affiliation: Master of Science of Fixed Prosthodontic department-Cairo University.

Name: Prof. Dr. Gihan El Naggar Rule: (Main Supervisor*)

*Responsible for implementation and allocation concealments.

* Data monitoring Affiliation: Professor of Fixed Prosthodontics- Faculty of Oral and Dental Medicine - Cairo University.

Name: Dr. Karim Abu Bakr Rule: (Co. Supervisor*) *Responsible for assignment of the patients in different groups during period of trial.

Affiliation: Lecturer of Fixed Prosthodontics - Faculty of Oral and Dental Medicine - Cairo University.

Supervisors direct and guide the practical work of the trial and give the final approval together with the EBD committee for the methodology of reporting the trial and for proceeding to publishing it later on.

5.b. Trial sponsor: Faculty of Oral and Dental Medicine, Cairo University, Egypt. 5.c. Role of trial sponsor: The trial sponsor will have no role in the design of this study and will have no role during its execution, analyses, interpretation of the data, or decision to submit results.

5.d. Steering committees:

1. Fixed Prosthodontics department Board: will review and approve the research plan and ensure that adequate methodology is carried out.
2. Research Plan Committee: To ensure that the trial satisfies the research plan of the Faculty and the department and to approve the methodological outcome.
3. Evidence Based Committee, Faculty of Oral and Dental Medicine - Cairo University, to ensure evidence based approval of the methodology and reporting of the trial.
4. Ethics Committee, Faculty of Oral and Dental Medicine - Cairo University: will ensure that the study meets the code of ethics of scientific research.
5. Higher Education and Research Committee.
6. Faculty Board.

II. Introduction 6.a. Background and rational 6.a.1. Background Endodontically treated teeth often show marked coronal mutilation,(1) which influence the structural integrity of such teeth and pose a higher risk of biomechanical failure than vital teeth.(2)

Traditionally those teeth are restored using post retained full coverage crowns.(3) Such treatment was thought to be the ideal way of restoring endodontically treated teeth while reinforcing the remaining tooth structure.(4) However, it was reported by many authors that placing a post can enhance the retention of the coronal restoration and the crown but at the same time carrying out the preparation for post insertion can weaken the remaining tooth structure, and hence increasing the risk of catastrophic tooth fracture.(5)

All-ceramic endocrowns are bonded to the tooth using adhesive resins creating strong bonds to the tooth structure resulting in strengthening effect and reducing the need for post and core.(6) various CAD/CAM materials can be used for the fabrication of endocrowns including lithium-disilicate reinforced glass-ceramics, feldspathic ceramics, in ceram alumina and in ceram spinell as well as hybrid ceramics and composites.(7)

6.a.2 Description of research question

Formulated question:

In patients with endodontically treated molar teeth requiring endocrown restorations, what are the clinical performance and the level of patient satisfaction of cerasmart endocrown versus lithium disilicate (e-max) ceramic endocrowns? 6.a.3 Justification for undertaking the trial: In 2016 Borgia et al. in their retrospective study to report the clinical performance of 11 endocrowns over a period of 9-18 years concluded that Endocrown being a conservative and aesthetic approach can be used to restore posterior endodontically treated teeth, mainly molars, with a very good biomechanical and functional performance, and very acceptable longevity. (22) Also the clinical performance of ceramic endocrowns showed a survival rate of 99 % and the success rate of 89.9 % in a 10 year retrospective study done by Bellflamme et al. 2017, where lithium disilicate (IPS Empress 2 or e-max) constituted 84.8 % of the functioning endocrowns while 12.1 % for polymer infiltrated ceramic (Vita Enamic) and only 3 % for artisanal indirect composite.(7)

However, lithium disilicate ceramics have disadvantages that may influence the outcome of the endocrowns, among which is the high stiffness and rigidity owing to the higher modulus of elasticity (67.2 GPa)(18) compared to natural dentin (18.6 GPa)(19) which may affect the marginal adaptation.(12) Moreover, high stress values will be induced with a detrimental effect on the biomechanical behavior of the restorative system when used to replace dentin.(20)

Rationale:

From a biomimetic point of view, the less brittle composite CAD/CAM blocks offer mechanical properties that are closely related to those of human dentin.(6) Nano ceramic material being more resilient and having lower stiffness and lower elastic modulus (12.1 GPa)(23) comparable to that of human dentin (18.6)(24) can act as a cushion and offer force absorption qualities thus reducing the stresses transferred to the adhesive junction.(25)

Benefits of the research to the patient:

Patient will receive a restoration with superior marginal adaptation and quality.

It will provide the patient with long-term predictable prosthetic outcome.

Benefits of the research to the clinician:

Practitioner will have the advantage to assess a new material that can be used in different situations for better marginal adaptation outcomes and bio integration.

It will improve patient's confidence with the dentist.

6.b. Explanation for choice of comparators: Ceramic material used for endocrown fabrication should be of acid etchable quality in order to obtain the necessary retention for such restoration through the adhesive cementation system.(15) thus lithium disilicate either machined or pressed seem to be the best restorative options in this case.(26)

In 2012 Biacchi and Basting reported that lithium disilicate ceramics possess a high bonding capacity to the dental structure which makes them the best restorative materials for endocrowns.(27)

Moreover lithium disilicates have been reported to offer high mechanical strength combined with exceptional esthetics which mimics greatly natural tooth appearance.(15) 7.a. Objectives: The aim of this study is to evaluate the clinical performance and patient satisfaction of new flexible ceramic material Cerasmart compared to lithium disilicate endocrowns.

7.b. Research hypothesis: Cerasmart endocrowns may have better clinical performance if compared with Lithium disilicate ceramic endocrown restorations.

8. Trial design: Randomized Clinical Trail (parallel group with 1:1 allocation ratio) A Superiority trial. III. A. Methods: Participants, interventions, and outcomes 9. Study setting: This study will be carried out on patients enrolled from the Outpatient clinic in fixed prosthodontics clinic, Faculty of Oral and Dental Medicine, Cairo University.

10. Eligibility criteria:

11. Interventions: 11.a. Main procedures: Methods

1. Patients collecting:

   (E.M) will select no of patients from outpatient clinic in fixed prosthodontic department clinic regarding previously mentioned inclusion and exclusion criteria.

   Suitable participants will be informed about the experimental trial and the possible complications that could occur during the period of this experiment. Each participant will be asked to sign informed consents, which will be provided in patient native language.
2. Tooth preparation and restoration placement:

(E.M) is responsible for all clinical procedure that will be conducted in this study

Pre-operative phase:

- Clinical records will be taken including history, clinical examination and clinical photographs

* Radiographs will be taken for the proposed abutments.
* Primary impressions will be taken and poured to obtain the study casts.

  1. st visit: (E.M) will call all selected participant before tooth preparation procedure for X-ray reviewing and pre-operative photographing using a digital camera also; primary impression will be taken using alginate impression material * for study cast analysis combined with suitable size stock tray**.
  2. nd visit: (Tooth preparation) After performing adequate disinfection and sterilization procedures for each instrument and tool that will be used in this trial, endocrown preparation will be carried out following the principles of endocrown preparation with a circumferential butt joint margin (of 1.5-2 mm thickness) with a reduction of at least 2 mm in the axial direction and a central retention cavity (of 3mm depth) making the coronal pulp chamber and the endodontic access cavity continuous. Walls less than 2 mm thick will be removed. 1-2 mm of Flowable composite resin base will be used to fill the undercuts. 2 observers will select visually the appropriate shade. Secondary impressions will be taken for each participant in each group using silicon rubber base impression material *** combined with suitable size tray Impressions will be removed from patient mouth after final setting and will be checked for accuracy

This will be followed by temporization using temporary filling material **** and will be left till the placement of endocrown in the next visit.

Impressions will be sent to the lab, which will be poured with extra hard stone material, after final setting of casts; it will be removed from the impression.

Casts will then be scanned using a scanning unit and then data will be saved on the computer.

Restoration fabrication:

Using Cerec in Lab software 4.2, a design of the desired e-max and cerasmart endocrowns will be planned in the form of a fully anatomical molar with a standardized proposal from the software this proposal will then be saved on the computer.

The e-max block as well as the cerasmart block will be fixed into its place in the wet milling machine, then the milling preview will be screened to check for any further adjustment, and finally an order will be given to the milling machine to mill the endocrowns.

3rd visit: Participants will be called again for final cementation. Temporary filling will be removed and abutments will be cleaned of any residues using pumice slurry ***** applied with bristle brush and rubber cup under water irrigation.

Proper isolation will be done before cementation then permanent resin cement ******will be used for luting of the endocrowns according to the manufacturer instructions. The patients will be requested to hold the endocrowns under occlusal compression until luting cement polymerization. After 5 minutes, excess cement will be removed.

Measuring of different outcomes will be in this visit for all patients. 11.b. Criteria for discontinuing interventions Conditions for discontinuing the prosthetic treatment include disappearance of the patient with loss of contact or patient's own request.

11.c. Strategies to improve adherence to intervention protocol: Face-to-Face adherence reminder session will take place in the initial visit. This session will include: the patient should be informed about the study steps and maintain oral hygiene. Subsequent sessions will occur at the follow-up visits. Participants will be asked about any problems they are having like pain, and oral hygiene.

11.d. Relevant concomitant care and interventions that are Permitted or prohibited during the trial: Motivation and maintenance of oral hygiene measures.

12. OUTCOMES

The following assessment surveys (clinical evaluations) will be carried out for both groups:

T1 = immediately after restoration delivery periapical radiograph. T2 = postoperatively: assessment of the restoration for patient satisfaction. The primary outcomes including retention, marginal adaptation, anatomic form, secondary caries, and surface texture will be examined using sharp explorer.

The secondary outcomes including modified gingival bleeding index and gingival periodontal index will be assessed and measured using periodontal explorer.

Both the primary as well as the secondary outcomes will be measured at baseline, after 1 month, then after 3 months and finally after 6 months (28) which will be enough for any color change or soft tissue response to take place.(29) Patients will be asked to give their restorations a grade out of 10 in order to indicate the level of their satisfaction.

All the grades of all the patients in both groups will be collected (for the alpha, bravo and Charlie) and the scores for the modified gingival index and the gingival periodontal index and aggregation will be done for the results.

For the clinical performance outcome, aggregates of all the alpha grades will be grouped as well as for the bravo and Charlie grades, then a percentage will be calculated for each grade.

For the soft tissue response outcome, the discrete scores will be gathered and grouped (0-4) for the modified gingival index and (0-5) for the gingival periodontal index and a percentage will be calculated for each group.

For the patient satisfaction outcome, the results will be grouped in five groups (0-2, 3-4, 5-6, 7-8 and 9-10) and a median will be drawn for each group.

13. Participant timeline:

The patient will be treated in visits designated as follows:

* Visit (1): Preoperative records, signing consents, clinical, radiographic examination and primary impression for diagnostic cast construction.
* Visit (2): Teeth preparation, secondary impression and temporary restorations.
* Visit (3): try in
* Visit (4): Placement and permanent cementation of the final restoration (endocrown) on the prepared tooth.

Assessment of clinical performance and patient satisfaction.

14. Sample size:

15. Recruitment: Patients fulfilling the inclusion criteria will be selected from the outpatient clinic of the fixed prosthodontics department - Cairo University.

Screening of patients will be carried out until the target population is reached.

III. B. Methods: Assignment of interventions 16. Allocation:

Patients grouping and allocations:

(E.G) will divide participants into two groups each (n=). Regarding restoration type, allocation will be done using software application and implementation will be carried out by (E.G) to insure validity of the trial (www.randomizer.com).

16.a. Sequence generation (E.G) will allocate participants into two groups with 1:1 allocation ratio by using computerized Sequence generation (www.randomizer.org). Simple randomization will be used.

16.b. Allocation concealments: (E.G) will write generated numbers by indispensable pen on large white paper sheet. The sheet will be folded eight times and saved inside opaque well sealed envelope in which the inner content cannot be seen by naked eyes.

16.c. Implementation: Each patient will select one of the envelopes that were previously well sealed and (A.K) will open the envelopes and assign the patients into the groups.

17. Blinding: Participants, operator, outcome assessor and statistical analyst will be blinded to avoid performance, detection and analysis bias. Only (E.G) and (A.K) will be aware of the allocated patients in each group and the specific type of intervention given to every patient.

(E.M) will be responsible for all experimental procedures and outcomes assessment.

III. C. Methods: data collection, management, and analysis Methods 18. Data collection methods: (E.M) will assess the outcomes of each group. Primary outcome: the two groups will be assessed using the modified United States public health service (USPHS) criteria as follows • Alpha (Excellent) ideal.

* Bravo (Acceptable) less than ideal but no modifications required
* Charlie (Acceptable but modifications needed) staining or other shade modifications required.

Secondary outcome: (patient satisfaction) of the two groups will be assessed using the Visual Analogue Scale (VAS) which is discrete and will be documented in chart including number of satisfied and unsatisfied.

Secondary outcome: soft tissue response will be assessed using Modified Gingival bleeding index MGI and Gingival Periodontal Index GPI which are discrete scores (0-4 and 0-3 respectively) and will be documented in chart.

Plans to promote participant retention & complete follow-up:

Telephone numbers and address of the patient included in the study will be recorded. All patients will be given a phone call and text message before the next appointment.

19. Data management: (A.K) will enter all data electronically. Patient files are to be stored in numerical order in a secured place.

20. Statistical methods: All Data will be collected, checked, revised, tabulated and entered into the computer. Quantitative variables from normal distribution will be expressed as mean and standard deviation (SD) values.

III. D. Monitoring:

21. Data monitoring The main supervisor is responsible for data monitoring if harms arise; (lost, deleted) in that case: back up will be asked from (E.M) to provide hard copy for the requested data.

22. Harms: Unintended adverse effects will be collected, assessed and reported if any happened.

23. Auditing: Auditing of the study design will be done by the evidence based committee - Faculty of Oral and Dental medicine - Cairo University.

IV. Ethics and dissemination 24. Research ethics approval This protocol and the template informed consent form will be reviewed by the Ethics Committee of Scientific Research - faculty of Oral and dental medicine - Cairo University.

25. Protocol amendments: Any modifications to the protocol which may impact on the conduct of the study, potential benefit of the patient or may affect patient safety, including changes of study objectives, study design, sample sizes, study procedures, or significant administrative aspects will require a formal amendment to the protocol. Such amendment will be agreed upon by the Council of the Department of fixed prosthodontics, Faculty of Oral and Dental Medicine, Cairo University.

26. Consent: Researcher will discuss the trial with all patients. Patients will then be able to have an informed discussion with the researcher. Researcher will obtain written consent from patients willing to participate in the trial. All consent forms will be in Arabic language (Appendix 1.1).

27. Confidentiality: All study-related information will be stored securely. All participants' information will be stored in locked file cabinets in areas with limited access. All data collection, process, and administrative forms will be identified by a coded ID [identification] number only to maintain participant confidentiality. All records that contain names or other personal identifiers will be stored separately from study records identified by code number. All local databases will be secured with password-protected access systems.

28. Declaration of interests: This trial is self-funded by the PhD student for the requirement PhD degree of fixed prosthodontics, Faculty of Oral and Dental Medicine Cairo University.

He does not have any conflict of interests with manufacturing companies, and is not a member of the Speaker's Panel of any company.

29. Access to data: The investigator and supervisors will be given access to the data sets. All data sets will be password protected. To ensure confidentiality, Participant study information will become confidentially.

30. Ancillary and post-trial care: All patients will be followed up until complete period study& patients' satisfactions occur. As any prosthetic treatment post insertion adjustment is necessary and in this trial recalls maintenance.

31. Dissemination policy:

* Study results will be published as partial fulfillment of the Requirements for PhD degree in fixed prosthodontics.
* Topics suggested for presentation or publication will be circulated to the authors.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of the patients from 15-60 years old.
2. Patients able physically and psychologically to tolerate conventional restorative procedures.
3. Patients with endodontically treated molars.
4. Patients with adequate root canal treatment with good apical seal.
5. Presence of teeth in opposite arch with normal occlusion.
6. Supra-gingival margin after preparation.
7. One wall defect cavity.
8. Patients willing to return for follow-up examinations and evaluation.

Exclusion Criteria:

1. Patients in the growth stage with partially erupted teeth.
2. Patients with poor oral hygiene and motivation.
3. Patients with parafunctional habits.
4. Patients with active periodontal or periapical disease.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Retention | 6 months
  Modified USPHS
  Primary outcome: the two groups will be assessed using the modified United States public health service (USPHS) criteria as follows
  * Alpha (Excellent) ideal.
  * Bravo (Acceptable) less than ideal but no modifications required
  * Charlie (Acceptable but modifications needed) staining or other shade modifications required.
  All the grades of all the patients in both groups will be collected (for the alpha, bravo and Charlie) and the scores for the modified gingival index and the gingival periodontal index and aggregation will be done for the results.
  For the clinical performance outcome, aggregates of all the alpha grades will be grouped as well as for the bravo and Charlie grades, then a percentage will be calculated for each grade.
Marginal adaptaion | 6 months
  Modified USPHS Primary outcome: the two groups will be assessed using the modified United States public health service (USPHS) criteria as follows
  * Alpha (Excellent) ideal.
  * Bravo (Acceptable) less than ideal but no modifications required
  * Charlie (Acceptable but modifications needed) staining or other shade modifications required.
  All the grades of all the patients in both groups will be collected (for the alpha, bravo and Charlie) and the scores for the modified gingival index and the gingival periodontal index and aggregation will be done for the results.
  For the clinical performance outcome, aggregates of all the alpha grades will be grouped as well as for the bravo and Charlie grades, then a percentage will be calculated for each grade.
Marginal discoloration | 6 months
  Modified USPHS
  Primary outcome: the two groups will be assessed using the modified United States public health service (USPHS) criteria as follows
  * Alpha (Excellent) ideal.
  * Bravo (Acceptable) less than ideal but no modifications required
  * Charlie (Acceptable but modifications needed) staining or other shade modifications required.
  All the grades of all the patients in both groups will be collected (for the alpha, bravo and Charlie) and the scores for the modified gingival index and the gingival periodontal index and aggregation will be done for the results.
  For the clinical performance outcome, aggregates of all the alpha grades will be grouped as well as for the bravo and Charlie grades, then a percentage will be calculated for each grade.
Anatomic form | 6 months
  Modified USPHS
  Primary outcome: the two groups will be assessed using the modified United States public health service (USPHS) criteria as follows
  * Alpha (Excellent) ideal.
  * Bravo (Acceptable) less than ideal but no modifications required
  * Charlie (Acceptable but modifications needed) staining or other shade modifications required.
  All the grades of all the patients in both groups will be collected (for the alpha, bravo and Charlie) and the scores for the modified gingival index and the gingival periodontal index and aggregation will be done for the results.
  For the clinical performance outcome, aggregates of all the alpha grades will be grouped as well as for the bravo and Charlie grades, then a percentage will be calculated for each grade.
Secomdary caries | 6 months
  Modified USPHS
  Primary outcome: the two groups will be assessed using the modified United States public health service (USPHS) criteria as follows
  * Alpha (Excellent) ideal.
  * Bravo (Acceptable) less than ideal but no modifications required
  * Charlie (Acceptable but modifications needed) staining or other shade modifications required.
  All the grades of all the patients in both groups will be collected (for the alpha, bravo and Charlie) and the scores for the modified gingival index and the gingival periodontal index and aggregation will be done for the results.
  For the clinical performance outcome, aggregates of all the alpha grades will be grouped as well as for the bravo and Charlie grades, then a percentage will be calculated for each grade.
Surface texture | 6 months
  Modified USPHS
Color match | 6 months
  Modified USPHS
  Primary outcome: the two groups will be assessed using the modified United States public health service (USPHS) criteria as follows
  * Alpha (Excellent) ideal.
  * Bravo (Acceptable) less than ideal but no modifications required
  * Charlie (Acceptable but modifications needed) staining or other shade modifications required.
  All the grades of all the patients in both groups will be collected (for the alpha, bravo and Charlie) and the scores for the modified gingival index and the gingival periodontal index and aggregation will be done for the results.
  For the clinical performance outcome, aggregates of all the alpha grades will be grouped as well as for the bravo and Charlie grades, then a percentage will be calculated for each grade.

SECONDARY OUTCOMES:
Modified Gingival bleeding index MGI | 6 months
  Modified Gingival bleeding index MGI:
  0 absence of inflammation
  1. mild inflammation
  2. moderate, bright surface inflammation ofgingival marginal or papillary
  3. mild inflammation in all portions of gingival marginal or papillary
  4. severe inflammation
  The secondary outcomes including modified gingival bleeding index and gingival periodontal index will be assessed and measured using periodontal explorer.
  For the soft tissue response outcome, the discrete scores will be gathered and grouped (0-4) for the modified gingival index
Modified Periodontal Index | 6 months
  Modified Periodontal Index:
  0 Tissue tightly adapted to the teeth Slight to moderate inflammation
  1. moderate inflammation completely encircle one or more teeth in a segment.
  2. Slight to moderate inflammation
  3. Marked inflammation indicated by loss of surface continuity
  For the soft tissue response outcome, the discrete scores will be gathered and grouped (0-3) for the gingival periodontal index and a percentage will be calculated for each group
Patient satisfaction | 6 months
  Visual Analogue Scale Patients will be asked to give their restorations a grade out of 10 in order to indicate the level of their satisfaction.
  For the patient satisfaction outcome, the results will be grouped in five groups (0-2, 3-4, 5-6, 7-8 and 9-10) and a median will be drawn for each group.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gihan El Nagar, Study Director — Professor, Fixed Prosthodontics department, Cairo University
Locations (1):
- Cairo University, Giza, Egypt

REFERENCES:
- [Background] Naumann M, Blankenstein F, Dietrich T. Survival of glass fibre reinforced composite post restorations after 2 years-an observational clinical study. J Dent. 2005 Apr;33(4):305-12. doi: 10.1016/j.jdent.2004.09.005. Epub 2004 Dec 10. PMID 15781138
- [Background] Guo J, Wang Z, Li X, Sun C, Gao E, Li H. A comparison of the fracture resistances of endodontically treated mandibular premolars restored with endocrowns and glass fiber post-core retained conventional crowns. J Adv Prosthodont. 2016 Dec;8(6):489-493. doi: 10.4047/jap.2016.8.6.489. Epub 2016 Dec 15. PMID 28018567
- [Background] Bitter K, Kielbassa AM. Post-endodontic restorations with adhesively luted fiber-reinforced composite post systems: a review. Am J Dent. 2007 Dec;20(6):353-60. PMID 18269124
- [Background] 4. Moradpoor H, Raissi S. Survival Rate of Endodontically Treated Teeth with Fiber Posts after Prosthodontic Restoration: A Study Review. Sch J Dent Sci. 2017;4(2):43-